CLINICAL TRIAL: NCT06238934
Title: Treatment of Knee Osteoarthritis With Bone Marrow Aspirate Matrix: Prospective, Randomized Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Traumatologia e Ortopedia (Other Government)
Responsible Party: Principal Investigator, Eduardo Branco de Sousa, Orthopaedic surgeon, Instituto Nacional de Traumatologia e Ortopedia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 74952423.1.0000.5273
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; knee; hyaluronic acid; bone marrow aspirate; bone marrow aspirate matrix
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Bone marrow aspirate matrix
  Interventions: Biological: Bone marrow aspirate matrix
- Group B (Active Comparator): Bone marrow aspirate
  Interventions: Biological: Bone marrow aspirate
- Group C (Active Comparator): Hyaluronic acid
  Interventions: Device: Hyaluronic acid

INTERVENTIONS:
Biological: Bone marrow aspirate matrix — Bone marrow aspirate * Hyaluronic acid
  Arms: Group A
Biological: Bone marrow aspirate — Bone marrow aspirate
  Arms: Group B
Device: Hyaluronic acid — Hyaluronic acid
  Arms: Group C

SUMMARY:
Knee osteoarthritis (KOA) first manifests itself as a molecular derangement followed by anatomical and/or physiological changes. Conservative treatment of osteoarthritis should be the first approach to patients with this disease. The interest in biological therapies, including viscosupplementation and cell therapy, involves the recent update in knowledge about the pathophysiology of OA and its natural history. The aim of the present study is to compare the clinical results of intra-articular hyaluronic acid infiltration (IHA), bone marrow aspirate (BMA) and BMA matrix in the treatment of knee osteoarthritis. The sample will consist of 90 patients with osteoarthritis of the knee followed up at the INTO, who will be divided into three groups: group A, treatment with BMA; group B, treatment with IHA ; and group C, treatment with BMA matrix. Patients will be submitted to clinical, subjective functional and radiographic evaluation by an observer independent of the one who applied the selected treatment, at moments before application and 3 months, 6 months and 12 months after application. We believe that treatment with BMA and the BMA matrix have a better effect in improving symptoms and for a longer period of time than treatment with hyaluronic acid.

ELIGIBILITY:
Inclusion Criteria:

Bilateral knee OA according to the American College of Rheumatology criteria Kellgren-Lawrence ≤ III in both knees Full range of movement (0 a 120°).

Exclusion Criteria:

1) history of trauma, infection or previous surgery in the affected limb two years before procedure (2)limb malalignment: varus> 10° or valgus >15° (3) corticosteroids 3 months before the procedure (4) viscosupplementation 12 months before procedure (5) inflammatory, rheumatological or autoimmune disease (6) body mass index >35 kg/m2 (7) use of immunosuppresors or anticoagulants (8) active tumor (9) haematological disorder (10) Hip OA > Tonnis grade 3 (11) history of transmissible disease (12) patients unable for positioning for the procedure (13) patients living outside Rio de Janeiro metropolitan area

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score | before infiltration, 1 month after first infiltration, three months, six months and one year after infiltration
Western Ontario and Mcmaster (WOMAC) score | before infiltration, 1 month after first infiltration, three months, six months and one year after infiltration
Visual analog scale for pain | before infiltration, 1 month after first infiltration, three months after infiltration, six months and one year after infiltration

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Traumatologia e Ortopedia, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No